CLINICAL TRIAL: NCT02851173
Title: Cognitive Enhancement Through Transcranial Laser Therapy
Acronym: LLLT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Andreana P. Haley, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-09-0018
Record Dates: First submitted 2016-07-27; First posted 2016-08-01 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Healthy Participants; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLLT (Experimental): Six weekly sessions of LLLT. The treatment will consist of applying light of a specific wavelength (1064 nm) using a laser diode supplied by Cell Gen Therapeutics, LLC (CG-5000 laser, HD Laser Center, Dallas, TX, USA). Each laser stimulation session will consist of total 8 min, with eight 1 min/cycle treatments alternating between two locations on the right forehead.
  Interventions: Device: LLLT
- Placebo (Active Comparator): The control group will undergo the same procedure as the treatment group, but will receive brief (5-s) stimulation to the intended site on the forehead, followed by 55 s of no stimulation, for each 1-min cycle. Thus the control group will receive approximately 1/12th of the cumulative energy density as the treatment group. This is sufficient to provide a brief sensation of slight heat (as active placebo) at the onset of each one-minute cycle, using a fraction of the energy received by the experimental group.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: LLLT — The treatment will consist of applying light of a specific wavelength (1064 nm) using a laser diode supplied by Cell Gen Therapeutics, LLC (CG-5000 laser, HD Laser Center, Dallas, TX, USA).
  Arms: LLLT
Device: Placebo — The treatment will consist of applying light of a specific wavelength (1064 nm) using a laser diode supplied by Cell Gen Therapeutics, LLC (CG-5000 laser, HD Laser Center, Dallas, TX, USA). However, the placebo group will receive approximately 1/12th of the cumulative energy density as the treatment group.
  Arms: Placebo

SUMMARY:
This is a mechanism-driven translational project to test the efficacy of transcranial low-level light/laser therapy (LLLT), for enhancing cognitive function in middle-aged and older adults and participants with Mild Cognitive Impairment.

DETAILED DESCRIPTION:
The goal of this project is to test the efficacy of LLLT to enhance neurocognitive function in middle-aged adults and examine the modulating influences of carotid atherosclerosis. The specific aims will be accomplished in a randomized controlled trial (RCT) by examining cognitive test performance and blood oxygen level-dependent (BOLD) response to a working memory task in middle-aged and older adults and participants with Mild Cognitive Impairment pre- and post- six-week long intervention of LLLT or placebo. In addition, the investigators will examine if carotid artery intima-media thickness (IMT) moderates the therapeutic effects of LLLT.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women, aged 45 and older
* Participants with Mild Cognitive Impairment

Exclusion Criteria:

* neurological disease (e.g., large vessel stroke, seizure disorder, Parkinson's disease, Alzheimer's disease, clinically significant traumatic brain injury with loss of consciousness > 30 minutes, multiple sclerosis, or brain infection/meningitis
* baseline IQ < 85 placing them below the average range of intellectual functioning
* major psychiatric illness (e.g., schizophrenia, bipolar disorder) or substance abuse (diagnosed abuse and/or previous hospitalization for substance abuse)
* severe cardiovascular disease (e.g., pacemaker), chronic obstructive pulmonary disease, liver or kidney disease, inflammatory illness

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-02-21 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Haley, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 641 participants were screened, 155 passed initial phone screening, 91 were enrolled and randomized.
Period: Overall Study
Arm/Group | LLLT | Placebo
Started | 44 | 47
Completed | 42 | 43
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LLLT | Placebo | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.4) | 64.4 (9.5) | 64.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 17 | 19 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 36 | 73
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 5 | 9 | 14
Psychomotor Vigilance Task (PVT) [Mean (Standard Deviation); unit: msec] — The psychomotor vigilance task (PVT) is a sustained-attention, reaction-timed task that measures the consistency with which subjects respond to a visual stimulus. Population: Missing data
  msec
    number analyzed (Participants) | 40 | 42 | 82
    (all) | 338.2 (96.8) | 342.8 (53.94) | 340.5 (77.4)

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Vigilance Task (PVT)
Description: The psychomotor vigilance task (PVT) is a sustained-attention, reaction-timed task that measures the consistency with which subjects respond to a visual stimulus.
Time Frame: Time 1 represents PVT performance (reaction time in msec) at baseline, Time 2 represents PVT performance (reaction time in msec) six weeks later.
Population: Cognitively unimpaired (CU) participants were analyzed separately from the Mild Cognitive Impairment (MCI) participants. One participant was missing data on T1 and 2 participants were missing data on T2 due to equipment failure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | LLLT | Placebo
Number analyzed (Participants) | 40 | 43
msec
  Time 1 CU: number analyzed (Participants) | 28 | 30
  Time 1 CU | 341.89 (47.8) | 344.09 (58.03)
  Time 2 CU: number analyzed (Participants) | 28 | 30
  Time 2 CU | 331.11 (62.85) | 330.75 (45.97)
  Time 1 MCI: number analyzed (Participants) | 12 | 13
  Time 1 MCI | 329.76 (165.87) | 339.81 (45.53)
  Time 2 MCI: number analyzed (Participants) | 11 | 13
  Time 2 MCI | 333.94 (139.73) | 321.19 (62.40)
Statistical Analysis 1: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. CU group; Test type: Other; p = 0.79, ANOVA
Statistical Analysis 2: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. MCI group; Test type: Other; p = 0.87, ANOVA
Statistical Analysis 3: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. CU group. 3 outliers removed, whose scores were outside 1.5 times the interquartile range; Test type: Other; p = 0.16, ANOVA

2. Secondary Outcome: Brain Blood Oxygen Level Dependent Response to Working Memory (2Back) Task
Description: The outcome represents a score on a scale - brain activation in response to a working memory task (t-statistic). The range is approximately -15 to +15. Positive scores reflect greater engagement of working memory brain regions and better performance.
Time Frame: T1 represents score at baseline; T2 represents follow-up score, 6 weeks later
Population: No data were collected on the secondary outcome variables from participants with Mild Cognitive Impairment (MCI) per study design as this task is too difficult for people with cognitive impairment. Two participants were missing T1 data due to equipment failure; 2 participants were missing T2 due to equipment failure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LLLT | Placebo
Number analyzed (Participants) | 28 | 30
score on a scale
  CU T1 Left middle frontal gyrus 1.: number analyzed (Participants) | 27 | 30
  CU T1 Left middle frontal gyrus 1. | 2.47 (2.59) | 3.00 (1.54)
  CU T2 Left middle frontal gyrus 1.: number analyzed (Participants) | 28 | 29
  CU T2 Left middle frontal gyrus 1. | 2.51 (2.40) | 3.39 (2.15)
  CU T1 Left medial frontal/superior frontal gyrus.: number analyzed (Participants) | 27 | 30
  CU T1 Left medial frontal/superior frontal gyrus. | 2.90 (2.22) | 2.67 (1.36)
  CU T2 Left medial frontal/superior frontal gyrus.: number analyzed (Participants) | 28 | 29
  CU T2 Left medial frontal/superior frontal gyrus. | 3.06 (2.17) | 2.89 (2.29)
  CU T1 Right superior parietal lobule.: number analyzed (Participants) | 27 | 30
  CU T1 Right superior parietal lobule. | 2.50 (2.47) | 2.81 (1.72)
  CU T2 Right superior parietal lobule.: number analyzed (Participants) | 28 | 29
  CU T2 Right superior parietal lobule. | 2.39 (2.96) | 2.86 (2.57)
  CU T1 Left inferior parietal lobule.: number analyzed (Participants) | 27 | 30
  CU T1 Left inferior parietal lobule. | 2.87 (2.39) | 3.46 (1.71)
  CU T2 Left inferior parietal lobule.: number analyzed (Participants) | 28 | 29
  CU T2 Left inferior parietal lobule. | 3.09 (2.71) | 3.36 (2.35)
  CU T1 Left middle frontal gyrus 2.: number analyzed (Participants) | 27 | 30
  CU T1 Left middle frontal gyrus 2. | 1.80 (2.11) | 2.02 (1.60)
  CU T2 Left middle frontal gyrus 2.: number analyzed (Participants) | 28 | 29
  CU T2 Left middle frontal gyrus 2. | 1.84 (1.72) | 2.14 (2.12)
  CU T1 Right superior frontal gyrus.: number analyzed (Participants) | 27 | 30
  CU T1 Right superior frontal gyrus. | 2.26 (2.36) | 2.50 (1.59)
  CU T2 Right superior frontal gyrus.: number analyzed (Participants) | 28 | 29
  CU T2 Right superior frontal gyrus. | 1.93 (2.15) | 2.85 (2.38)
  CU T1 Right middle frontal gyrus.: number analyzed (Participants) | 27 | 30
  CU T1 Right middle frontal gyrus. | 3.09 (2.90) | 3.51 (2.04)
  CU T2 Right middle frontal gyrus.: number analyzed (Participants) | 28 | 29
  CU T2 Right middle frontal gyrus. | 3.31 (2.80) | 3.89 (2.86)
  CU T1 Right inferior frontal gyrus.: number analyzed (Participants) | 27 | 30
  CU T1 Right inferior frontal gyrus. | 0.72 (2.00) | 1.19 (2.13)
  CU T2 Right inferior frontal gyrus.: number analyzed (Participants) | 28 | 29
  CU T2 Right inferior frontal gyrus. | 1.14 (2.13) | 1.27 (2.47)
Statistical Analysis 1: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Left middle frontal gyrus 1; Test type: Other; p = 0.22, ANOVA
Statistical Analysis 2: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Left medial frontal/superior frontal gyrus; Test type: Other; p = 0.69, ANOVA
Statistical Analysis 3: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Right superior parietal lobule; Test type: Other; p = 0.25, ANOVA
Statistical Analysis 4: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Left inferior parietal lobule; Test type: Other; p = 0.86, ANOVA
Statistical Analysis 5: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Left middle frontal gyrus 2; Test type: Other; p = 0.28, ANOVA
Statistical Analysis 6: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Right superior frontal gyrus; Test type: Other; p = 0.12, ANOVA
Statistical Analysis 7: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. Right middle frontal gyrus; Test type: Other; p = 0.26, ANOVA
Statistical Analysis 8: Comparison: LLLT vs Placebo; The contract of interest was the Time x Treatment Group interaction. Right inferior frontal gyrus; Test type: Other; p = 0.83, ANOVA
Statistical Analysis 9: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Left middle frontal gyrus 1; Test type: Other; p = 0.55, ANOVA
Statistical Analysis 10: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Left medial frontal/superior frontal gyrus; Test type: Other; p = 0.76, ANOVA
Statistical Analysis 11: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Right superior parietal lobule; Test type: Other; p = 0.38, ANOVA
Statistical Analysis 12: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Left inferior parietal lobule; Test type: Other; p = 0.93, ANOVA
Statistical Analysis 13: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Left middle frontal gyrus 2; Test type: Other; p = 0.41, ANOVA
Statistical Analysis 14: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Right superior frontal gyrus; Test type: Other; p = 0.06, ANOVA
Statistical Analysis 15: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Right middle frontal gyrus; Test type: Other; p = 0.18, ANOVA
Statistical Analysis 16: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy). Right inferior frontal gyrus; Test type: Other; p = 0.84, ANOVA

3. Secondary Outcome: Working Memory (2 Back Task)
Description: 2Back task performance (%Correct)
Time Frame: T1 represents 2back % Correct at baseline; T2 represents 2back % Correct 6 weeks later
Population: No data were collected on the secondary outcome variables from participants with Mild Cognitive Impairment (MCI) per study design as this task is generally too difficult for patients with cognitive impairment. Data were missing on 7 participants at T1 and 9 participants on T2 due to equipment failure.
Measure: Mean (Standard Deviation); unit: % correct responses of total responses
Arm/Group | LLLT | Placebo
Number analyzed (Participants) | 27 | 25
% correct responses of total responses
  CU %Correct T1 | 73.93 (14.57) | 73.54 (13.48)
  CU %Correct T2: number analyzed (Participants) | 26 | 24
  CU %Correct T2 | 77.17 (14.97) | 79.59 (13.01)
Statistical Analysis 1: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction; Test type: Other; p = 0.53, ANOVA
Statistical Analysis 2: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction. In this sub-group analysis, we performed a sub-population analysis (N=36), including only participants who performed the 2Back task to criterion (>50% accuracy); Test type: Other; p = 0.74, ANOVA

4. Secondary Outcome: Working Memory (2 Back Task)
Description: 2Back task performance (Reaction Time in msec)
Time Frame: T1 represents 2back Reaction Time (RT) in msec at baseline; T2 represents Reaction Time (RT) in msec 6 weeks later
Population: No data were collected on the secondary outcome variables from participants with Mild Cognitive Impairment (MCI) per study design as this task is generally too difficult for people with cognitive impairment. Data were missing on 10 participants at T1 and 13 participants on T2 due to equipment failure.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | LLLT | Placebo
Number analyzed (Participants) | 26 | 23
msec
  CU RT T1 | 1289.19 (225.72) | 1173.98 (268.44)
  CU RT T2: number analyzed (Participants) | 23 | 23
  CU RT T2 | 1202.89 (261.49) | 1035.05 (271.38)
Statistical Analysis 1: Comparison: LLLT vs Placebo; The contrast of interest was the Time x Treatment Group interaction; Test type: Other; p = 0.72, ANOVA
Statistical Analysis 2: Comparison: LLLT vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.97, ANOVA

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected for the duration of the study (12 weeks)
Arm/Group | LLLT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/47
Other Adverse Events (participants affected / at risk) | 0/44 | 2/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LLLT (N=44) | Placebo (N=47)
pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — 24 hours post screening blood draw, participant reported floating pain (started in the arm, moved to back, and "haunches")
headache (Nervous system disorders) | 0 (0) | 1 (1) — participant reported headaches, judged to be related to an unrelated medical condition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02851173/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT02851173/SAP_001.pdf